CLINICAL TRIAL: NCT01625780
Title: A New Approach to Ilio-inguinal Nerve Blocks: 3-layer Injection vs Conventional Ultrasound-guided Single-shot Approach
Brief Title: Comparing Ilioinguinal Single-shot and Three-layer Blocks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not a significant difference in outcomes between groups
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00027444
Record Dates: First submitted 2012-04-12; First posted 2012-06-21 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2016-10

CONDITIONS: Ilioinguinal Nerve Block; Local Anesthesia; Post-operative Analgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group: 3-layer block (Experimental): Patients in this group will receive the 3-layer ilioinguinal nerve block.
  Interventions: Procedure: 3-layer block
- Control: single-shot block (Active Comparator): Patients in this group will receive a standard, single-shot ilioinguinal nerve block.
  Interventions: Procedure: Single-shot block

INTERVENTIONS:
Procedure: 3-layer block — 0.3 mL/kg of 0.25% bupivacaine (one injection in each layer) will be delivered by the "3-layer" method using a standard 20-gauge block needle.
  Arms: Study group: 3-layer block
Procedure: Single-shot block — 0.3 mL/kg of 0.25% bupivacaine will be delivered by the standard, single-shot method using a 20-gauge block needle.
  Arms: Control: single-shot block

SUMMARY:
Ilio-inguinal nerve blocks have a long history of efficacy in treatment of post-operative pain following inguinal surgery. Several anatomic studies have shown that the nerves supplying the inguinal area have a certain degree of variability with respect to their location between the internal and external oblique layers of the anterior abdominal wall. Furthermore, the standard single-shot approach to ilio-inguinal nerve blocks has a significant incidence of unintended femoral nerve block, which can impair patients' ability to walk after surgery. The investigators are proposing a new approach to the ilio-inguinal nerve block, which divides the total dose of local anesthetic into 3 equal parts, injecting each 1/3 into different layers of the anterior abdominal wall and sub-cutaneously. The investigators intend to show that this new technique, the Tsui approach, provides equal analgesia to the standard single-shot ultrasound-guided ilio-inguinal nerve block, while being faster to perform and having a lower incidence of unintended femoral nerve blockade. Patients under age 10 who are scheduled for elective inguinal surgery (hydrocele repair, orchidopexy, and inguinal hernia repair), who have already consented to an ilio-inguinal nerve block that is commonly placed for this type of procedure, will be approached to participate in this study. No increased risk is anticipated for these patients, as both ultrasound-guided and blind techniques are equally well-accepted in the literature for this type of block, and in addition there are few vascular or neural structures in this anatomical area (just medial and inferior to the anterior superior iliac spine) that may be damaged. Follow-up will be limited to an assessment of pain scores in the PACU post-operatively and any unintended femoral nerve blockade in post-PACU. This will not delay their hospital discharge as these are same-day surgery patients.

DETAILED DESCRIPTION:
Project Summary Rationale - The conventional technique for performing an ilio-inguinal nerve block involves a single shot of local anesthetic (usually 0.3 mL/kg of 0.25% bupivacaine) in the transversus abdominis plane of the anterior abdominal wall. Using a blind technique (also known as "fascial click"), a blunted needle (20 gauge) is placed 1 cm medial and 1 cm inferior to the anterior superior iliac spine (ASIS), and directed downward perpendicular to the skin surface until two distinct "pops" are felt, corresponding to the external and internal oblique fascial layers. The entire volume of local anesthetic is then deposited in this plane. Success with this technique ranges from 35-75% in the literature (1-3). Studies have shown that volumes as low as 0.075 mL/kg of 0.25% levobupivacaine have provided equal analgesia to 0.2 mL/kg for up to 4 hours post-operatively when ultrasound guidance is used to ensure placement of local anesthetic near the ilio-inguinal and/or ilio-hypogastric nerves (4), resulting in a 100% success rate for this block.

We are proposing a technique that will deliver 1/3 of the total dose of local anesthetic (0.3 mL/kg of 0.25% bupivacaine) for each layer of the lower anterior abdominal wall. Due to the anatomic variability of the course of the ilio-inguinal and ilio-hypogastric nerves, we believe that the placement of 0.1 mL/kg in each of the external oblique, internal oblique, and transversus abdominis layers will improve the success of the "fascial click" approach without the need for ultrasound guidance. In addition, the ilio-inguinal nerve block has a known complication of unintended femoral nerve block. The incidence of femoral nerve block varies from 4.5% to 9% (5); in fact, one randomized controlled trial of ilio-inguinal nerve block for inguinal hernia repair in adults had to be stopped prior to completion due to patient harm (falls, etc) from femoral nerve blockade (6). We propose that a 3-layer technique will have a lower incidence of unintended femoral nerve block as compared to the conventional single-shot technique.

For inguinal surgery (orchidopexy, inguinal hernia repair, or hydrocele repair), both the ilio-inguinal and ilio-hypogastric nerves need to be blocked. The ilio-inguinal nerve arises from L1 and follows the inguinal canal to innervate the medial aspect of the thigh, anterior scrotum or labia. The ilio-hypogastric nerve has an anterior cutaneous branch the runs at the level of the ASIS, providing innervation to the skin and subcutaneous tissues of the inguinal region. For orchidopexy surgery, additional local anesthetic may be needed if the scrotal incision is towards the apex of the scrotum (posterior - perineal nerve vs anterolateral - genito-femoral nerve) rather than on the anterior aspect.

Study Goals and Objectives Primary Objective - To introduce a new technique of IHN/IIN blocks that is equianalgesic to the single-shot technique without requiring ultrasound guidance.

Secondary Objective - To introduce a technique that has a lower incidence of unintended femoral nerve block.

Study Design Randomized controlled trial comparing two groups: single-shot group (0.3 mL/kg of 0.25% bupivacaine placed 1 cm medial to the ASIS following two "pops" via the fascial click method), and the three-shot (TS) group, where 1/3 of the total dose above is deposited in each of the 3 layers (external and internal oblique, transversus abdominis). In the TS group, 0.1 mL/kg of 0.25% bupivacaine will be injected per layer.

Methods After IRB approval, ASA I-II children presenting for inguinal surgery (orchidopexy, inguinal hernia, or hydrocele repair) whose parents have already given consent for an ilio-inguinal nerve block, will be approached to participate in this study. Written informed consent will be obtained from parents, while verbal assent will be obtained from children where appropriate. Exclusion criteria include patient or parental refusal, local anesthetic allergy, or contraindication to ilio-inguinal nerve block.

The ilio-inguinal nerve blocks will be performed by the attending anesthesiologist who is responsible for the child's anesthetic. Each child will be premedicated with 20 mg/kg of oral acetaminophen. Induction of anesthesia will be intravenous (propofol and remifentanil) or via facemask (oxygen and sevoflurane) according to the discretion of the attending anesthetist. Following placement of intravenous access and laryngeal mask airway, anesthesia will be maintained with 1 MAC (minimum alveolar concentration) of sevoflurane in air/O2 with spontaneous ventilation. Intraoperative monitoring will include heart rate, electrocardiogram, oxygen saturation, non-invasive arterial blood pressure, and end-tidal carbon dioxide, oxygen concentration, and anesthetic agent.

A SonoSite ultrasound unit (SonoSite M-Turbo, Bothell, WA, USA) and a SLAx 13-6 MHz linear hockey stick probe will be used to document the placement of the local anesthetic and the relevant anatomical structures. The study investigators will turn the screen away from the attending anesthesiologist performing the block and will save 'before' and 'after' images of the block onto a USB stick via the ultrasound machine. The attending anesthesiologist will sterilize the area with chlorhexidine solution and locate the ASIS. Using a blunted 20 gauge needle, they will place the needle approximately one finger's-breadth medial to the ASIS and insert perpendicular to the skin until 2 pops are felt. If the patient has been randomized to the single-shot group, following negative aspiration, all of the local anesthetic (0.3 mL/kg of 0.25% bupivacaine) will be injected here. A screen shot of local anesthetic spread will then be saved through the ultrasound machine onto a USB stick. If the patient has been randomized to the three-shot (TS) group, following negative aspiration, one third of the local anesthetic (0.1 mL/kg of 0.25% bupivacaine) will be injected here, then pulled back one "pop" to the next layer where another third of the local anesthetic will be injected. The final third of the local anesthetic dose will be injected subcutaneously in a skin wheal medial to the ASIS. Again, a screen shot of local anesthetic spread will be saved via the ultrasound machine to a USB stick. The USB stick will be password-protected using only consecutive numbers to identify the patients. The investigator who will later review the screen shots from the ultrasound will thus be blinded from patient allocation.

Following block placement, the surgeon may prep and drape the patient in preparation for the surgical procedure. Baseline heart rate and arterial blood pressure will be noted following skin incision. An increase in heart rate or arterial blood pressure greater than 20% from baseline will be treated with rescue analgesia (fentanyl 1 mcg/kg IV). For orchidopexy, additional local anesthetic (0.1 mL/kg 0.25% bupivacaine) will be used for local infiltration of the scrotal incision.

Post-operatively, analgesia will be recorded by trained pediatric nurses in the post-anesthetic care unit (PACU) using the FLACC pain scale for young children or non-verbal patients, and using the Wong-Baker Faces Pain Score for older children. Both are rated on a scale of 0-10. Any score greater than 6 will be treated with morphine 0.05 mg/kg IV, up to 2 doses, 15 minutes apart. PACU nurses will also note any quadriceps weakness, indicating an unintended femoral nerve block. Following discharge from PACU, the patients will continue to be monitored for pain scores in day surgery area for up to 4 hours post-operatively. No follow-up is planned beyond discharge from day surgery.

Studies have shown that a blind, single shot technique for ilio-inguinal nerve blocks has a success rate of 35-75% (1-3). For the purposes of our study, we will use a value of 60% efficacy for the single-shot technique. We hypothesize that a 3-shot technique will have an efficacy of 90%, based on studies showing 100% efficacy for single-shot ultrasound-guided technique (4), and 94% efficacy in a similar study (7). For a power of 0.8, alpha 0.05, we calculate a sample size of 32 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II children aged 0-16 presenting for inguinal surgery (inguinal hernia, hydrocele repair, or orchidopexy)

Exclusion Criteria:

* Patient or parent refusal to participate in study, local anesthetic allergy, or any other contraindication to ilio-inguinal nerve block.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Time to completion of block for equal analgesia (intraoperative or post-operative need for rescue analgesia) | From identification of needle insertion site to end of injection of local anesthetic (single shot blocks are typically completed within 5 minutes)
  Time (in seconds/minutes) taken to achieve a satisfactory ilioinguinal nerve block will be recorded.

SECONDARY OUTCOMES:
Time to onset of block | When maximal nerve block is achieved (after approximately 20 minutes for single-shot blocks)
  Time taken to achieve effective nerve block will be recorded.
Change in heart rate upon surgical incision | At the moment the skin incision is made (varies; intra-operative)
  Patient heart rate will be recorded at the moment the surgical incision is made.

CONTACTS AND LOCATIONS:
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Langer JC, Shandling B, Rosenberg M. Intraoperative bupivacaine during outpatient hernia repair in children: a randomized double blind trial. J Pediatr Surg. 1987 Mar;22(3):267-70. doi: 10.1016/s0022-3468(87)80344-5. PMID 3550031
- [Background] Splinter WM, Bass J, Komocar L. Regional anaesthesia for hernia repair in children: local vs caudal anaesthesia. Can J Anaesth. 1995 Mar;42(3):197-200. doi: 10.1007/BF03010675. PMID 7743568
- [Background] Dalens B, Ecoffey C, Joly A, Giaufre E, Gustafsson U, Huledal G, Larsson LE. Pharmacokinetics and analgesic effect of ropivacaine following ilioinguinal/iliohypogastric nerve block in children. Paediatr Anaesth. 2001 Jul;11(4):415-20. doi: 10.1046/j.1460-9592.2001.00691.x. PMID 11442857
- [Background] Willschke H, Bosenberg A, Marhofer P, Johnston S, Kettner S, Eichenberger U, Wanzel O, Kapral S. Ultrasonographic-guided ilioinguinal/iliohypogastric nerve block in pediatric anesthesia: what is the optimal volume? Anesth Analg. 2006 Jun;102(6):1680-4. doi: 10.1213/01.ane.0000217196.34354.5a. PMID 16717308
- [Background] Lim SL, Ng Sb A, Tan GM. Ilioinguinal and iliohypogastric nerve block revisited: single shot versus double shot technique for hernia repair in children. Paediatr Anaesth. 2002 Mar;12(3):255-60. doi: 10.1046/j.1460-9592.2002.00832.x. PMID 11903940
- [Background] Walker S, Orlikowski C. A randomised study of ilio-inguinal nerve blocks following inguinal hernia repair: a stopped randomised controlled trial. Int J Surg. 2008 Feb;6(1):23-7. doi: 10.1016/j.ijsu.2007.10.003. Epub 2007 Oct 24. PMID 18053781
- [Background] Willschke H, Marhofer P, Bosenberg A, Johnston S, Wanzel O, Cox SG, Sitzwohl C, Kapral S. Ultrasonography for ilioinguinal/iliohypogastric nerve blocks in children. Br J Anaesth. 2005 Aug;95(2):226-30. doi: 10.1093/bja/aei157. Epub 2005 May 27. PMID 15923270